CLINICAL TRIAL: NCT06836388
Title: Ultrasound-Guided Bougie Insertion Technique and Conventional Method in Difficult Intubation: A Randomized Controlled Study
Brief Title: Using Ultrasound for Bougie Insertion in Difficult Airway Management
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Mohammed Gaber Saad (Other)
Responsible Party: Sponsor-Investigator, Mohammed Gaber Saad, Lcturer of anesthesia, intensive care and pain medicine, Al-Azhar University
Organization: Al-Azhar University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Anesth-.0434/2024 Med research
Record Dates: First submitted 2025-01-28; First posted 2025-02-20 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-01

CONDITIONS: Difficult Airway
Keywords: ultrasound; Difficult airways; Bougie

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Group A: Ultrasound-guided bougie insertion (Active Comparator): the ultrasound will be used to provide a real-life observation of the bougie advancement into the trachea to confirm its correct placement.
  Interventions: Procedure: ultrasound guided bougie insertion
- Group B: Conventional bougie insertion (Placebo Comparator): using the conventional method for bougie insertion
  Interventions: Procedure: Conventional methods for bougie insertion

INTERVENTIONS:
Procedure: ultrasound guided bougie insertion — The anesthesiologist will use a high-frequency linear ultrasound probe at the level of the suprasternal notch to identify the tracheal rings. The probe will then be moved cephalad and placed over the cricothyroid membrane to visualize the vocal folds in the transverse view with the patient in the supine position. Using a C-mac laryngoscope, the intubator will assess the difficulty of visualization using the Cormack Lehan score; if the score is three or more, the bougie will be gently inserted with the curved tip anteriorly into the trachea and assess the real-time visualization of the bougie on the ultrasound screen as a linear echogenic structure moving through the hypoechoic lumen of the trachea then the tube will railed on the bougie and connected to the capnograph for endotracheal positioning confirmation when the square waveform will be maintained for five breaths.
  Arms: Group A: Ultrasound-guided bougie insertion
Procedure: Conventional methods for bougie insertion — The anesthesiologist will perform the bougie insertion using a C-mac laryngoscope, and he will assess the difficulty of visualization using the Cormack Lehan score; if the score is three or more, the bougie will be gently inserted with the curved tip anteriorly into the trachea while feeling the tracheal clicks as a sign of correct its placement, the intubator will advance it gently till feel resistance then withdraw 2-3 centimeters. If the depth of the bougie reaches 30 centimeters from the angle of the mouth without feeling the resistance, the bougie will be removed and reinserted. Then, the tube will be railed on the bougie and connected to the capnograph for endotracheal positioning confirmation when the square waveform is maintained for five breaths.
  Arms: Group B: Conventional bougie insertion

SUMMARY:
Difficult airway management remains one of the biggest challenges in anesthesia practice. The Gum elastic bougie, an intubation tool, is frequently used to facilitate intubation in difficult situations. Recently, ultrasound-guided airway management has been used as a potential method to improve the intubation process. This study aims to compare the efficacy of ultrasound-guided bougie insertion with the conventional method regarding the duration of endotracheal tube (ETT) insertion and the number of attempts required in a difficult intubation population.

The goal of this clinical trial is to learn if using ultrasound during bougie insertion in difficult airway patients will improve the success rate and reduce the time of insertion. The main questions it aims to answer are:

Does using ultrasound reduce the number of insertion attempts? Does using ultrasound reduce the duration of bougie insertion?

Researchers will compare the ultrasound-guided technique to the conventional bougie insertion method. They will also assess both groups' hemodynamic parameters during and after the procedure and the success rate from the first trial.

ELIGIBILITY:
Inclusion Criteria:

* Adults aged 15 -75 years.
* Elective surgical operation.
* ASA (American Society of Anesthesiologists) physical status I-III.
* Predicted difficult airway.

Exclusion Criteria:

* Emergency intubations.
* Patients with contraindications to the use of bougie.
* Patients with a known allergy to local anesthetics or ultrasound gel.
* Pregnancy.
* Craniofacial anomaly
* Patients with obstructive sleep apnea
* BMI > 35.
* Patient with gastroesophageal reflux disease.

Ages: 15 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2024-09-23 (Actual); Primary Completion 2025-03-30 (Actual); Study Completion 2025-04-30 (Estimated)

PRIMARY OUTCOMES:
Duration of bougie insertion. | during the insertion of bougie
  the time in seconds from the start of the bougie insertion to successful ETT placement
Number of attempts required for successful bougie insertion | during the insertion of bougie
  As each separate insertion of the bougie: if the bougie cannot visualized by the ultrasound in (group A) OR if the depth of the bougie reaches 30 centimeters depth from the angle of the mouth without feeling the resistance in (group B), the bougie will be withdrawn and reinserted again.

SECONDARY OUTCOMES:
Systolic and daistolic blood pressure changes during intubation | T1: 5 minutes before induction of anesthesia. T2: 5 minutes after tube positioning confirmation. T3:15 minutes after tube positioning confirmation
  The systolic blood pressure in mmHg at T1, T2 and T3. The diastolic blood pressure in mmHg at T1, T2 and T3
Success rate of the first attempt | during the insertion of bougie
  Count the cases in which the insertion of bougie was confirmed from the first insertion trial.
Hemodynamic changes during intubation | T1: 5 minutes before induction of anesthesia. T2: 5 minutes after tube positioning confirmation. T3:15 minutes after tube positioning confirmation
  The systolic blood pressure in mmHg at T1, T2 and T3. The diastolic blood pressure in mmHg at T1, T2 and T3 Heart rate per minute at T1, T2 and T3
Heart rate during the procedure | Pulse rate per minute T1: 5 minutes before induction of anesthesia. T2: 5 minutes after tube positioning confirmation. T3:15 minutes after tube positioning confirmation
  The pulse rate per minute will be observed and documented at T1, T2 and T3

CONTACTS AND LOCATIONS:
Locations (1):
- Faculity of medicine - Al-Azhar University hospitals, Cairo, Cairo Governorate, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Huan C, Pan H, Fu S, Xu W, Gao Q, Wang X, Gao S, Chen C, Liu X. Characterization and evolution of the coronavirus porcine epidemic diarrhoea virus HLJBY isolated in China. Transbound Emerg Dis. 2020 Jan;67(1):65-79. doi: 10.1111/tbed.13321. Epub 2019 Aug 22. PMID 31381232
- [Background] Moore CL, Copel JA. Point-of-care ultrasonography. N Engl J Med. 2011 Feb 24;364(8):749-57. doi: 10.1056/NEJMra0909487. No abstract available. PMID 21345104
- [Background] Driver BE, Prekker ME, Klein LR, Reardon RF, Miner JR, Fagerstrom ET, Cleghorn MR, McGill JW, Cole JB. Effect of Use of a Bougie vs Endotracheal Tube and Stylet on First-Attempt Intubation Success Among Patients With Difficult Airways Undergoing Emergency Intubation: A Randomized Clinical Trial. JAMA. 2018 Jun 5;319(21):2179-2189. doi: 10.1001/jama.2018.6496. PMID 29800096
- [Background] Kristensen MS. Ultrasonography in the management of the airway. Acta Anaesthesiol Scand. 2011 Nov;55(10):1155-73. doi: 10.1111/j.1399-6576.2011.02518.x. Epub 2011 Sep 7. PMID 22092121